CLINICAL TRIAL: NCT03455764
Title: A Phase I/II Study of MCS110 With BRAF/MEK Inhibition in Patients With Melanoma After Progression on BRAF/MEK Inhibition
Brief Title: MCS110 With BRAF/MEK Inhibition in Patients With Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Elizabeth Buchbinder, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-656
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 1] (Experimental): * MCS110 2.5mg/kg will be administered intravenously every 3 weeks.
  * Dabrafenib 150mg is given orally every 12 hours.
  * Trametinib 2mg is given orally daily
  Interventions: Drug: MCS110; Drug: Dabrafenib; Drug: Trametinib
- MCS110 + Trametinib + Dabrafenib [Phase 2] (Experimental): * MCS110 will be administered intravenously every 3 weeks. The Dosage will be determined by the DLT of Phase 1
  * Dabrafenib 150mg is given orally every 12 hours.
  * Trametinib 2mg is given orally daily
  Interventions: Drug: MCS110; Drug: Dabrafenib; Drug: Trametinib
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level -1] (Experimental): * MCS110 1.25 mg/kg was administered intravenously every 3 weeks.
  * Dabrafenib 150mg is given orally every 12 hours.
  * Trametinib 2mg is given orally daily
  Interventions: Drug: MCS110; Drug: Dabrafenib; Drug: Trametinib
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 2] (Experimental): * MCS110 5mg/kg was administered intravenously every 3 weeks.
  * Dabrafenib 150mg is given orally every 12 hours.
  * Trametinib 2mg is given orally daily
  Interventions: Drug: MCS110; Drug: Dabrafenib; Drug: Trametinib
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 3] (Experimental): * MCS110 10mg/kg was administered intravenously every 3 weeks.
  * Dabrafenib 150mg is given orally every 12 hours.
  * Trametinib 2mg is given orally daily
  Interventions: Drug: MCS110; Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: MCS110 — MCS110 is a colony-stimulating factor-1 (CSF-1) inhibitor. It is a human monoclonal antibody which binds CSF-1.
Drug: Dabrafenib — Dabrafenib attack different proteins that promote the growth of cancerous cells
  Other Names: Tafinlar
Drug: Trametinib — Trametinib attack different proteins that promote the growth of cancerous cells
  Other Names: Mekinist

SUMMARY:
This research study is studying a combination of targeted therapies as a possible treatment for advanced melanoma that was found to have a BRAF V600E or BRAF V600K genetic mutation.

The interventions involved in this study are:

* MCS110
* Dabrafenib
* Trametinib

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial. A Phase I clinical trial tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved MSC110 as a treatment for any disease.

The FDA has approved dabrafenib and trametinib as treatment options for this disease.

Dabrafenib and trametinib attack different proteins that promote the growth of cancerous cells. These two treatments work in cancers with a mutation in the BRAF gene which alters a protein signaling pathway in cancer cells. The BRAF mutation status will be confirmed during this trial by review or procedure in order to make sure this clinical trial is right for the participant. Dabrafenib is a BRAF inhibitor that works by preventing altered BRAF proteins from stimulating the growth of the melanoma cancer cells. Trametinib works by blocking a protein related to BRAF called MEK that has been known to stimulate cells that also promote melanoma growth. In order to participate in the study, the participant disease needs to be tested positive for a mutation (a permanent change in the DNA sequence of a gene) of the BRAF gene that belongs to a class of genes known as oncogenes. When mutated, oncogenes have the potential to cause normal cells to become cancerous. Once the BRAF gene is mutated, the normal functioning of the BRAF protein may be changed. It is normal for patients with a BRAF mutation to receive these types of inhibitor therapies at some point in their treatment.

MCS110 is a colony-stimulating factor-1 (CSF-1) inhibitor. It is a human monoclonal antibody which binds CSF-1. A monoclonal antibody is a type of protein made in the laboratory that can locate and bind to substances in the body, including tumor cells. MCS110 is being developed as a treatment for patients with advanced cancer.

In this research study, the investigators are adding MCS110 to the treatment with dabrafenib and trametinib at the time when the participant's disease is growing despite these medications. The hope is that MCS110 will enhance how the cancer will respond to dabrafenib and trametinib and overcome any resistance to these medications that has developed. In previous laboratory studies performed by treating melanoma cancer cells with a CSF-1R (CSF-1 Receptor which interacts with the CSF-1 protien) inhibitor and a BRAF inhibitor, it was found that the CSF-1R inhibitor was successful in increasing efficacy.

ELIGIBILITY:
Inclusion Criteria:

* For enrollment to the phase I portion: participants must have a histologically confirmed melanoma with a BRAF V600E or BRAF V600K mutation (identified via NextGen sequencing using the DFCI/BWH OncoPanel or any CLIA-certified method) that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective.
* For enrollment to the phase II portion: participants must have a histologically confirmed melanoma with a BRAF V600E or BRAF V600K mutation (identified via NextGen sequencing using the DFCI/BWH OncoPanel or any CLIA-certified method) and have had progression of disease on prior BRAF and MEK inhibitor therapy.
* Participants enrolling to the phase I portion of the trial must have evaluable or measurable disease.
* Participants enrolling to the phase II portion of the trial must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Age ≥ 18 years. As no dosing or adverse event data are currently available in participants < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
* ECOG performance status 0 - 2 (see Appendix A).
* Life expectancy of greater than 8 weeks.
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/uL
  * Platelets ≥ 100 K/uL
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN
  * Serum creatinine ≤ 1.5 × institutional ULN
  * PT-INR ≤ 1.5 × institutional ULN (for participants on anticoagulation therapy, ≤ 1.5 × their baseline value)
  * aPTT ≤ 1.5 × institutional ULN (for participants on anticoagulation therapy, ≤ 1.5 × their baseline value)
* Participants must have a left ventricular ejection fraction (LVEF) ≥ 50%.
* Participants must have a QTc of ≤ 470 msec for females and ≤ 450 for males on the screening EKG.
* The effects of MCS110, trametinib and dabrafenib on the developing human fetus are unknown. For this reason and because anti-cancer agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months after the last dose of MCS110. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of MCS110 administration. Highly Effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
  * Double-barrier contraception: condom and occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/cream/suppository).
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must have archival tumor tissue available. Participants without archival tissue may be enrolled at the discretion of the principal investigator.
* All prior anti-cancer treatment-related toxicities (except alopecia and laboratory values as listed on Table 1) must be ≤ Grade 1 according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.0; NCI, 2009) at the time of randomization

Exclusion Criteria:

* Participants who have had chemotherapy, radiotherapy, biologic therapy, major surgery, or another investigational agent within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Previous BRAF/MEK inhibitor use is allowed with no washout period for the phase I and II portions.
* Participants who have not recovered to ≤ CTCAE grade 1 or baseline from toxicity as a result of previous cancer treatment prior to entering the study (with the exception of alopecia and peripheral neuropathy which can be ≤ grade 2).
* For enrollment to the phase II portion: participants who have not received prior BRAF or MEK inhibitor therapy.
* Participants with known untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with a history of brain metastases that have been treated, are no longer taking corticosteroids, and have been stable on imaging for ≥ 4 weeks following the last date of treatment are permitted.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MCS110, dabrafenib, or trametinib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because MCS110, dabrafenib and trametinib are anti-cancer agents with the potential for teratogenic or abortifacient effects. Pregnancy status will be verified at various points in the trial and a serum pregnancy test will be required. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MCS110, dabrafenib or trametinib, breastfeeding should be discontinued if the mother is treated with MCS110, dabrafenib or trametinib.
* Participants with a known history of HIV are ineligible because of the potential for pharmacokinetic interactions with MCS110, dabrafenib, and trametinib with antiretroviral agents. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Participants with a personal or family history of long QT syndrome.
* Participants with a history of a second primary malignancy. Exceptions include: patients with a history of malignancies that were treated curatively and have not recurred within 3 years prior to study entry; resected basal and squamous cell carcinomas of the skin, and completely resected carcinoma in situ of any type.
* Participants with impairment of GI function or GI disease that may significantly alter the absorption of dabrafenib and trametinib in the opinion of the treating investigator (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* Participants who are unable to swallow or retain oral medication.
* Participants that require co-administration of strong or moderate CYP3A inhibitors, as these medications may alter dabrafenib and trametinib concentrations.
* Participants who require treatment with medications that are strong or moderate CYP3A inducers, as these medications may alter the concentration of trametinib.
* Participants with evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration.
* Participants with a history of or current evidence of retinal vein occlusion or retinal pigment epithelial detachment.
* Participants taking corticosteroids (≥ 10 mg of prednisone or equivalent). Exceptions may be discussed with the Overall PI on a case by case basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth I Buchbinder, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from September 2018 to July 2019.
Pre-assignment Details: Phase 2 never enrolled any patients because the company stopped development of the drug after the 6 patients were enrolled to the phase 1 portion. No further patients were enrolled to either arm after that.
Groups:
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 1]: MCS110 2.5 mg/kg was administered intravenously every 3 weeks. Dabrafenib 150mg is given orally every 12 hours. Trametinib 2mg was given orally daily.
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level -1]: MCS110 1.25 mg/kg was administered intravenously every 3 weeks. Dabrafenib 150mg is given orally every 12 hours. Trametinib 2mg was given orally daily.
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 2]: MCS110 5 mg/kg was administered intravenously every 3 weeks. Dabrafenib 150mg is given orally every 12 hours. Trametinib 2mg was given orally daily.
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 3]: MCS110 10 mg/kg was administered intravenously every 3 weeks. Dabrafenib 150mg is given orally every 12 hours. Trametinib 2mg was given orally daily.
- MCS110 + Trametinib + Dabrafenib [Phase 2]: MCS110 at recommended phase 2 dose level was administered intravenously every 3 weeks.
  Dabrafenib 150mg is given orally every 12 hours. Trametinib 2mg was given orally daily.
Period: Overall Study
Arm/Group | MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 1] | MCS110+ Trametinib + Dabrafenib [Phase I Dose Level -1] | MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 2] | MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 3] | MCS110 + Trametinib + Dabrafenib [Phase 2]
Started | 6 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 4 | 0 | 0 | 0 | 0
Not completed — On Treatment | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Zero patients were enrolled in the Phase 2 portion of this study.
Groups:
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 1]: MCS110 2.5 mg/kg was administered intravenously every 3 weeks. Dabrafenib 150mg was given orally every 12 hours. Trametinib 2mg was given orally daily.
- MCS110 + Trametinib + Dabrafenib [Phase 2]: MCS110 at recommended phase 2 dose level was administered intravenously every 3 weeks.
  Dabrafenib 150mg was given orally every 12 hours. Trametinib 2mg was given orally daily.
- Total: Total of all reporting groups
Arm/Group | MCS110+ Trametinib + Dabrafenib [Phase I Dose Level 1] | MCS110 + Trametinib + Dabrafenib [Phase 2] | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (17.1) |  | 53.7 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 3 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 6 |  | 6
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 6 |  | 6
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT) [Phase I]
Description: A DLT was defined as an adverse event that (a) was possibly, probably, or definitely related to the study medication regimen and (b) experienced during the first cycle of treatment, and (c) met any of the following criteria: ≥ Grade 3 non-hematological toxicity; grade 3 thrombocytopenia with clinically significant bleeding; grade 4 thrombocytopenia; ≥ grade 3 febrile neutropenia; grade 4 anemia; holding of any study medication due to toxicity for a period of greater than 8 consecutive days or two separate periods of any duration during the first cycle, any other significant toxicity deemed by the principal investigator to be dose limiting.
Time Frame: Participants were followed up to 21 days.
Population: The study was terminated before Phase 2 was initiated.
Measure: Count of Participants; unit: Participants
Groups:
- MCS110+ Trametinib + Dabrafenib: * For Phase 1 MCS110 2.5mg/kg will be administered intravenously every 3 weeks.
  * Dabrafenib 150mg is given orally every 12 hours.
  * Trametinib 2mg is given orally daily
Arm/Group | MCS110+ Trametinib + Dabrafenib
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Maximum Tolerated Dose of MCS110 [Phase I]
Description: The trial used 3+3 design to determine maximum tolerated dose (MTD), escalating on 0/3 or 1/6 DLTs, and de-escalating if two DLTs were encountered. See subsequent primary outcome measure for the DLT definition. MTD was the highest dose level at which 0/3 or 1/6 subjects experienced a DLT.
Time Frame: Participants were followed up to 21 days.
Measure: Number; unit: mg/kg
Arm/Group | MCS110+ Trametinib + Dabrafenib
Number analyzed (Participants) | 6
mg/kg | 2.5

3. Secondary Outcome: Overall Response Rate (ORR) [Phase I]
Description: ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Participants were followed up to 30 months.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | MCS110+ Trametinib + Dabrafenib
Number analyzed (Participants) | 6
percentage of participants | 16.7 [1 to 58]

4. Secondary Outcome: Median Progression Free Survival [Phase I]
Description: PFS is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anticancer therapy. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: Participants were followed up to 30 months.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | MCS110+ Trametinib + Dabrafenib
Number analyzed (Participants) | 6
months | 2.3 [1.3 to NA] — Insufficient number progressed during the time of observation.

5. Post Hoc Outcome: Grade 3 Adverse Events Rate
Description: Grade 3 adverse event (AE) rate was defined as the proportion of patients who experienced grade 3 adverse events based on Common Terminology Criteria for Adverse Events (CTCAE) version 4 (see standard source vocabulary as per AE module). Descriptions of severity (grade) are dependent on AE type with a scale of 1 (least severe) to 5. Please refer to https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm
  Per their definitions:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL).
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: Participants were followed up to 30 months.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | MCS110+ Trametinib + Dabrafenib
Number analyzed (Participants) | 6
proportion of participants | 0.83 [0.42 to 0.99]

6. Post Hoc Outcome: Median Overall Survival (OS)
Description: OS based on Kaplan-Meier method is defined as the time from registration to death due to any cause, or censored at date last known alive.
Time Frame: Participants were followed up to 30 months.
Population: Zero patients were enrolled in the Phase 2 portion of the study.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | MCS110+ Trametinib + Dabrafenib
Number analyzed (Participants) | 6
months | 5.3 [3.4 to NA] — Insufficient number died during the time of observation.

ADVERSE EVENTS:
Time Frame: Participants were followed up to 30 months.
Description: A serious adverse event is any adverse event during this study that results in one of the following outcomes: death; hospitalization for greater than 24 hours; prolonging an existing inpatient hospitalization; a life-threatening experience (that is, immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; considered significant by the investigator for any other reason. All other remaining adverse events will be considered as other adverse event.
Groups:
- MCS110+ Trametinib + Dabrafenib [Phase I Dose Level I]: * For Phase 1 MCS110 2.5mg/kg will be administered intravenously every 3 weeks.
  * Dabrafenib 150mg is given orally every 12 hours.
  * Trametinib 2mg is given orally daily
- MCS110 + Trametinib + Dabrafenib Phase 2: * MCS110 will be administered intravenously every 3 weeks. The Dosage will be determine by the DLT of Phase 1
  * Dabrafenib 150mg is given orally every 12 hours.
  * Trametinib 2mg is given orally daily
Arm/Group | MCS110+ Trametinib + Dabrafenib [Phase I Dose Level I] | MCS110 + Trametinib + Dabrafenib Phase 2
All-Cause Mortality (participants affected / at risk) | 3/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCS110+ Trametinib + Dabrafenib [Phase I Dose Level I] (N=6) | MCS110 + Trametinib + Dabrafenib Phase 2 (N=0)
Alkaline phosphatase increased (Investigations) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MCS110+ Trametinib + Dabrafenib [Phase I Dose Level I] (N=6) | MCS110 + Trametinib + Dabrafenib Phase 2 (N=0)
Anemia (Blood and lymphatic system disorders) | 4 | NA
Pericardial effusion (Cardiac disorders) | 1 | NA
Hypothyroidism (Endocrine disorders) | 1 | NA
Blurred vision (Eye disorders) | 1 | NA
Conjunctivitis (Eye disorders) | 1 | NA
Watering eyes (Eye disorders) | 1 | NA
Eye disorders - Other, specify (Eye disorders) | 2 | NA
Abdominal pain (Gastrointestinal disorders) | 2 | NA
Constipation (Gastrointestinal disorders) | 2 | NA
Diarrhea (Gastrointestinal disorders) | 4 | NA
Nausea (Gastrointestinal disorders) | 4 | NA
Oral hemorrhage (Gastrointestinal disorders) | 1 | NA
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | NA
Vomiting (Gastrointestinal disorders) | 4 | NA
Chills (General disorders) | 4 | NA
Edema limbs (General disorders) | 1 | NA
Fatigue (General disorders) | 3 | NA
Fever (General disorders) | 5 | NA
Flu like symptoms (General disorders) | 2 | NA
Infusion related reaction (General disorders) | 2 | NA
Malaise (General disorders) | 1 | NA
Pain (General disorders) | 1 | NA
Infections and infestations - Other, specify (Infections and infestations) | 1 | NA
Alanine aminotransferase increased (Investigations) | 2 | NA
Alkaline phosphatase increased (Investigations) | 3 | NA
Aspartate aminotransferase increased (Investigations) | 6 | NA
CPK increased (Investigations) | 5 | NA
Creatinine increased (Investigations) | 2 | NA
GGT increased (Investigations) | 1 | NA
Lipase increased (Investigations) | 1 | NA
Neutrophil count decreased (Investigations) | 1 | NA
Platelet count decreased (Investigations) | 1 | NA
Weight gain (Investigations) | 1 | NA
Weight loss (Investigations) | 2 | NA
White blood cell decreased (Investigations) | 2 | NA
Investigations - Other, specify (Investigations) | 1 | NA
Anorexia (Metabolism and nutrition disorders) | 3 | NA
Dehydration (Metabolism and nutrition disorders) | 3 | NA
Hypercalcemia (Metabolism and nutrition disorders) | 1 | NA
Hyperkalemia (Metabolism and nutrition disorders) | 1 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | NA
Hypocalcemia (Metabolism and nutrition disorders) | 1 | NA
Hypokalemia (Metabolism and nutrition disorders) | 2 | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | NA
Hyponatremia (Metabolism and nutrition disorders) | 2 | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | NA
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Dizziness (Nervous system disorders) | 2 | NA
Headache (Nervous system disorders) | 3 | NA
Memory impairment (Nervous system disorders) | 1 | NA
Paresthesia (Nervous system disorders) | 1 | NA
Syncope (Nervous system disorders) | 1 | NA
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | NA
Insomnia (Psychiatric disorders) | 1 | NA
Acute kidney injury (Renal and urinary disorders) | 1 | NA
Urinary frequency (Renal and urinary disorders) | 1 | NA
Urine discoloration (Renal and urinary disorders) | 1 | NA
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | NA
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | NA
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | NA
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | NA
Hot flashes (Vascular disorders) | 1 | NA

LIMITATIONS AND CAVEATS:
Early termination resulted from the drug manufacturer's decision to stop drug development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03455764/Prot_SAP_000.pdf